CLINICAL TRIAL: NCT07056010
Title: Efficacy and Safety of Minimally-invasive Curative Gastrectomy and D2+PAND Lymphadenectomy for Gastric Cancer Patients With Para-aortic Lymph Node (PAN) Metastasis After Conversion Immunochemotherapy
Brief Title: Efficacy and Safety of Minimally Invasive D2+PAND Gastrectomy for Gastric Cancer With PAN Metastasis After Conversion Immunochemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Xu, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL-D2PAND
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients will undergo curative minimally invasive gastrectomy with D2+PAND (Experimental)
  Interventions: Procedure: curative minimally invasive gastrectomy with D2+PAND lymphadenectomy

INTERVENTIONS:
Procedure: curative minimally invasive gastrectomy with D2+PAND lymphadenectomy — Thirty patients with HER2-negative gastric adenocarcinoma or gastroesophageal junction (GEJ) cancer, presenting with PAN metastasis (No. 16 lymph nodes ≥10 mm), will be enrolled. Participants will receive four cycles of conversion immunochemotherapy with a PD-1 inhibitor (Serplulimab) combined with the SOX chemotherapy regimen (oxaliplatin and S-1). After completion of conversion therapy, patients will undergo curative minimally invasive (laparoscopic or robotic) gastrectomy with D2+PAND lymphadenectomy.

SUMMARY:
This is a prospective, open-label, single-center, Phase II clinical trial. Thirty patients with HER2-negative gastric adenocarcinoma or gastroesophageal junction (GEJ) cancer, presenting with PAN metastasis (No. 16 lymph nodes ≥10 mm), will be enrolled. Participants will receive four cycles of conversion immunochemotherapy with a PD-1 inhibitor (Serplulimab) combined with the SOX chemotherapy regimen (oxaliplatin and S-1). After completion of conversion therapy, patients will undergo curative minimally invasive (laparoscopic or robotic) gastrectomy with D2+PAND lymphadenectomy

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, regardless of gender.

  * Histologically confirmed gastric cancer or gastroesophageal junction (GEJ) cancer that has received neoadjuvant therapy, with pathology confirming it is predominantly adenocarcinoma. For GEJ cancer, only Siewert Type III and Siewert Type II cases that do not require combined thoracotomy are eligible.
  * Tumor stage confirmed as cStage IV （ para-aortic lymph node enlargement without other distant metastatic factors）, suitable for curative R0 resection, as determined by an evaluation by a gastrointestinal surgeon and a radiologic technician prior to enrollment. The patient consented to conversion therapy followed by radical surgical resection, with no surgical contraindications confirmed by the attending surgeon.
  * No. 16 lymph nodes ≥10 mm
  * Subject must be previously untreated with systemic treatment; Subject that received neoadjuvant chemotherapy with recurrence >6 months from completion of therapy are permitted;
  * Expected survival of ≥6 months.
  * Measurable tumor lesions as defined by RECIST v1.1 criteria (see Attachment 1).
  * Preoperative ECOG performance status score (see Attachment 2) of 0 or 1.
  * Good cardiac function, capable of undergoing a curative resection. If there are clinical indications, patients with underlying ischemic, valvular heart disease, or other serious heart conditions should undergo preoperative assessment by a cardiologist.
  * Normal major organ function, with the following laboratory criteria:
  * Absolute neutrophil count (ANC) ≥ 1.2 x 10^9/L in the absence of granulocyte colony-stimulating factor use within the past 14 days.
  * Platelet count ≥ 100 x 10^9/L in the absence of blood transfusion within the past 14 days.
  * Hemoglobin > 8 g/dL in the absence of blood transfusion or erythropoietin use within the past 14 days.
  * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN); if total bilirubin > 1.5 × ULN but direct bilirubin ≤ ULN, inclusion is permitted.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.
  * Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by the Cockcroft-Gault formula) ≥ 60 mL/min.
  * Coagulation function defined by international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN.
  * Normal thyroid function, defined by thyroid-stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, patients with normal total T3 (or FT3) and FT4 levels may still be eligible.
  * Normal range for myocardial enzyme profile (patients with isolated laboratory abnormalities deemed clinically insignificant by the investigator may still be included).
  * Thyroid function tests (TSH, FT3/FT4) within normal limits or with minor clinically insignificant abnormalities.
  * Weight ≥ 40 kg (inclusive) or BMI > 18.5.
  * The participant has read, understood, and signed the informed consent form.

Exclusion Criteria:

* Patients with a history of (within the past 5 years) or current active malignancies. However, patients with cured localized tumors, such as basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, in situ prostate cancer, in situ cervical cancer, in situ breast cancer, stage I lung cancer, stage I colorectal cancer, etc., are eligible.

  * A history of upper abdominal surgery (except for laparoscopic cholecystectomy).
  * A history of gastric resection, endoscopic mucosal resection (EMR), or endoscopic submucosal dissection (ESD).
  * Patients requiring surgery for other diseases concurrently.
  * Emergency surgery performed due to complications of gastric cancer (e.g., bleeding, obstruction, or perforation).
  * Patients preparing for or with a history of organ or bone marrow transplantation.
  * Blood transfusion within 2 weeks prior to surgery or a history of bleeding disorders, or any severe bleeding event (grade 3 or above according to CTCAE 4.0) occurring within 4 weeks prior to surgery.
  * Coagulation disorders or bleeding tendencies (INR > 1.5 without anticoagulant use); patients receiving anticoagulants or vitamin K antagonists, such as warfarin, heparin, or similar agents. Low-dose warfarin (1 mg oral daily) or low-dose aspirin (≤100 mg daily) may be allowed for preventive purposes, provided the prothrombin time international normalized ratio (INR) is ≤ 1.5.
  * History of thromboembolic events (e.g., stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within 6 months prior to screening. Patients with venous thrombosis caused by prior chemotherapy and deemed healed by the investigator are excluded.
  * Myocardial infarction, poorly controlled arrhythmias (including QTc interval > 450 ms for males and > 470 ms for females) within 6 months prior to surgery. QTc interval should be calculated using the Fridericia formula.
  * NYHA class III or IV heart failure, or left ventricular ejection fraction (LVEF) < 50% as per echocardiogram.
  * Pulmonary dysfunction with FEV1 < 50% of predicted value.
  * Urinary protein ≥++ on routine urinalysis, confirmed by 24-hour urinary protein quantification > 1.0 g.
  * Clinically symptomatic pleural effusion or ascites requiring clinical intervention.
  * Human immunodeficiency virus (HIV) infection.
  * Active pulmonary tuberculosis.
  * Chronic non-healing wounds or fractures with incomplete healing.
  * History of interstitial lung disease, pneumoconiosis, radiation-induced pneumonitis, drug-induced pneumonitis, or severe pulmonary dysfunction that may interfere with the detection or management of potential drug-related pulmonary toxicity.
  * Known active or suspected autoimmune diseases, except those in stable condition at enrollment and without the need for systemic immunosuppressive therapy.
  * Severe chronic autoimmune diseases, such as systemic lupus erythematosus, inflammatory bowel diseases (e.g., ulcerative colitis, Crohn's disease), chronic diarrhea syndromes (e.g., irritable bowel syndrome), sarcoidosis, or tuberculosis. Active hepatitis B or C or HIV infections. Non-severe autoimmune conditions, such as controlled psoriasis, dermatitis, or arthritis, are eligible. Patients with hepatitis B virus (HBV) with a viral load < 500 copies/ml may be included.
  * Patients who require systemic corticosteroid treatment (> 10 mg/day prednisone equivalent) or other immunosuppressive drugs within 14 days prior to surgery or during the study period. However, the following are allowed for inclusion: patients without active autoimmune diseases may use topical or inhaled steroids or adrenal hormone replacement therapy with a dose ≤ 10 mg/day prednisone equivalent.
  * Patients who have an active infection requiring systemic antibiotic treatment within 14 days prior to surgery (excluding those receiving prophylactic antibiotics for conditions like urinary tract infections or chronic obstructive pulmonary disease).
  * Patients who have received live vaccines within 28 days prior to surgery; seasonal influenza vaccination with inactivated viral vaccines is excluded.
  * Patients currently enrolled in another clinical trial involving surgery-related treatments.
  * Patients with a history of alcoholism, drug abuse, or substance misuse. Patients who have stopped drinking alcohol are eligible.
  * Patients who do not comply with medical instructions, fail to follow prescribed medication regimens, or have incomplete data that could impact the assessment of efficacy or safety.
  * Pregnant or breastfeeding female patients.
  * Patients with conditions that may increase the risks of participating in the study or with other severe, acute, or chronic diseases deemed by the investigator to be unsuitable for participation.
  * Other situations determined by the investigator that make the patient unsuitable for this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2028-11-25 (Estimated)

PRIMARY OUTCOMES:
postoperative complications within 30 days after surgery | 30 days after surgery
  Early Postoperative Complications: Complications occurring within 30 days post-surgery (number of participants with treatment-related adverse events as assessed by CTCAE v4.0)

SECONDARY OUTCOMES:
Neoadjuvant treatment efficacy | 2 weeks after surgery
  R0 resection rate after neoadjuvant therapy
TRG | 2 weeks after surgery
  Tumor Regression Grade
pCR | 2 weeks after surgery
  pathological Complete Response

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical Unviersity, Nanjing, Jiangsu, China